CLINICAL TRIAL: NCT07065110
Title: A Single-center, Double-blind, Randomized, Parallel-group, Placebo-controlled Study to Evaluate the Superiority of Peroral Sodium Hyaluronate to Placebo in Improving the Skin Hydration
Brief Title: The Effect of Peroral Sodium Hyaluronate on the Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contipro Pharma a.s. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AICE24_II
Record Dates: First submitted 2025-06-12; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Skin Conditions
Keywords: skin; hydration
MeSH Terms: conditions — Skin Diseases | interventions — Blood Specimen Collection; xanthan gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA gel group (Experimental): Participants obtained altogether 3 flasks with 500 mL of SH60, SH120 solution. They took 15 mL of the SH60 or SH120 supplements (experimental groups) once daily in the morning before breakfast for 3 months.
  Interventions: Diagnostic Test: Blood draw for the laboratory assessment; Dietary Supplement: Skin test panel; Dietary Supplement: HA gel
- Xanthan gum group (Placebo Comparator): Participants obtained altogether 3 flasks of placebo solution. They took 15 mL of placebo solution (control group) once daily in the morning before breakfast for 3 months.
  Interventions: Diagnostic Test: Blood draw for the laboratory assessment; Dietary Supplement: Skin test panel; Dietary Supplement: Xanthan gum

INTERVENTIONS:
Diagnostic Test: Blood draw for the laboratory assessment — Blood draw for testing of metabolics.
Dietary Supplement: Skin test panel — Testing of improving the skin hydration and other skin-related parameters.
  Other Names: Skin condition testing
Dietary Supplement: HA gel — Participants obtained altogether 3 flasks with 500ml of SH60, SH 120 solution. They tooj 15 ml of the SH60 or SH120 aupplements (experimental group) once daily in the morning before breakfast for 3 months.
  Arms: HA gel group
Dietary Supplement: Xanthan gum — Participants obtained altogether 3 flasks of placebo solution. They took 15 mL of placebo solution (control group) once daily in the morning before breakfast for 3 months.
  Arms: Xanthan gum group

SUMMARY:
A single-center, double-blind, randomized, parallel-group, placebo-controlled study to evaluate the superiority of peroral sodium hyaluronate to placebo in improving the skin hydration and other skin-related parameters.

DETAILED DESCRIPTION:
Study type:

* Single-center, randomized, placebo-controlled, double-blind, parallel-group study.
* Participants will be stratified based on their sex (males/females) and age (young 18-39 years and old 40-60 years, max difference in median age between males and females 2 years), and randomly assigned to receive either the SH dietary supplements (lower concentration, daily dose 60 mg (SH60); and higher concentration, daily dose 120 mg (SH120)) or placebo in a 1:1:1 ratio.
* The study will follow a superiority framework, aiming to demonstrate that the SH60 and SH120 dietary supplements are superior to placebo in improving facial skin hydration.
* This study is a parallel-group trial: The three groups of participants (SH60/SH120/placebo group) will receive the treatments and will be assessed for their outcomes at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects
* Skin type: Caucasian, Fitzpatrick I-III
* Sex: male and female
* Age: 18 - 60 years.
* No acute or chronic skin diseases affecting the face or volar forearm.
* No acute or chronic gastrointestinal diseases.
* Willing to keep their standard facial skincare routine and avoid any new products or procedures affecting facial or volar forearm skin during the study period.
* Willing to avoid excessive UV exposure (tanning beds, excessive sunbathing) during the study period.
* Willing to avoid longer stays in significantly different climates (will be assessed on a case-by-case basis)
* Willing to avoid taking other dietary supplements containing SH

Exclusion Criteria:

* Subjects with known allergies to any ingredients in the dietary supplement.
* Pregnant or lactating individuals.
* Significant facial skin conditions or disorders.
* Acute or chronic disease affecting the skin or gastrointestinal system.
* Subjects currently using topical or oral medications affecting the gastrointestinal system or the skin.
* Subjects who are taking or has taken diet pills or supplements containing SH within the past 3 months.
* Subjects who are taking or has taken oral antibiotics in the last 3 months.
* Subjects with diabetes mellitus
* Subjects with increased bleeding tendency, poor superficial veins in the antecubital fossa, and those with a fear of blood draws that makes blood draw impossible

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Change in skin hydration | 0, 1, 2 , 3 months
  * Measurement site: forehead, volar forearm
  * Measurement time points: 0, 1, 2, 3 months
  * Measurement site: cheek
  * Measurement time points: 0, 1, 2 months
  * Measurement device: Corneometer CM 825
  * Parameter unit: AU (arbitrary unit)
  * Number of measurements at each time point: at least 5
  * Outcome measure: Change from baseline
  * Method of analysis:
    * Mean, standard deviation and confidence intervals will be calculated.
    * Normality of the data distribution will be assessed.
    * Comparison between HA group and placebo group will be assessed using independent sample T-test or Mann-Whitney U test as a nonparametric alternative.

SECONDARY OUTCOMES:
Change in TEWL | 0, 1, 2, 3 months
  * Measurement site: forehead, cheek
  * Measurement time points: 0 (baseline), 1, 2, 3 months
  * Measurement device: Tewameter TM 300
  * Parameter unit: AU (arbitrary unit)
  * Number of measurements at each time point: at least 10
  * Outcome measure: Change from baseline
  * Method of analysis:
    * Mean, standard deviation and confidence intervals will be calculated.
    * Normality of the data distribution will be assessed.
    * Comparison between HA group and placebo group will be assessed using independent sample T-test or Mann-Whitney U test as a nonparametric alternative.
Change in skin elasticity | 0, 1, 2, 3 months
  * Measurement site: forehead, cheek
  * Measurement time points: 0, 1, 2, 3 months
  * Measurement device: Cutometer MPA 580
  * Parameter unit: AU (arbitrary unit)
  * Number of measurements at each time point: at least 1
  * Outcome measure: Change from baseline
  * Method of analysis:
    * Mean, standard deviation and confidence intervals will be calculated.
    * Normality of the data distribution will be assessed.
    * Comparison between HA group and placebo group will be assessed using independent sample T-test or Mann-Whitney U test as a nonparametric alternative.
Change in wrinkle depth | 0, 1, 2, 3 months
  * Measurement site: crow´s feet area
  * Measurement time points: 0, 1, 2, 3 months
  * Measurement device: Primos Lite
  * Parameter unit: mm
  * Number of measurements at each time point: at least 3
  * Outcome measure: Change from baseline
  * Method of analysis:
    * Mean, standard deviation and confidence intervals will be calculated.
    * Normality of the data distribution will be assessed.
    * Comparison between HA group and placebo group will be assessed using independent sample T-test or Mann-Whitney U test as a nonparametric alternative.

CONTACTS AND LOCATIONS:
Locations (1):
- Contipro a.s., Ústí nad Orlicí, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doleckova I, Kusnierik P, Berka V, Simek M, Matejkova I, Prokopec F, Ovesna P. Oral sodium hyaluronate improves skin hydration, barrier function and signs of aging: a randomized, double-blind, placebo-controlled trial in 150 healthy adults. Sci Rep. 2025 Dec 20. doi: 10.1038/s41598-025-32758-5. Online ahead of print. PMID 41422283